CLINICAL TRIAL: NCT02754453
Title: An Evaluation of the Efficacy of a Group Treatment Intervention for Weight Regain After Bariatric Surgery-A Pilot Project
Brief Title: Weight Regain Study After Bariatric Surgery-A Pilot Project
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-129
Record Dates: First submitted 2013-09-25; First posted 2016-04-28 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-02

CONDITIONS: Behavioral; Activity; Weight Loss
Keywords: Weight Regain; Group Treatment; Weight Loss
MeSH Terms: conditions — Behavior; Motor Activity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Behavioral (Other)
  Interventions: Behavioral: Behavioral lifestyle intervention

INTERVENTIONS:
Behavioral: Behavioral lifestyle intervention — 20 session lifestyle behavioral intervention with the goal of altering diet and physical activity and decreasing problematic behaviors associated with weight regain and session behavioral intervention addressing increasing physical activity, improving adherence to dietary recommendations and altering problematic eating behaviors.

SUMMARY:
There are three different phases to this study:

1. Screening phase to determine if you are eligible to participate in the study.
2. Study phase, which will entail diet and activity, exercise and then finally self monitoring goals.
3. End of treatment phase where you will be asked to complete questionnaires.

DETAILED DESCRIPTION:
The purpose of this study is to determine the feasibility of a group treatment program for individuals experiencing weight regain after bariatric surgery and to evaluate the effectiveness of the group treatment program. There is little information on programs to assist patients who experience weight regain after bariatric surgery. This treatment program will focus on behavioral changes and activity.

ELIGIBILITY:
Inclusion Criteria:

* Weight regain post-RYGB of at least 5 kg since reaching their weight nadir.
* Male or Female age 18 - 65.
* Undergone RYGB 12 - 36 month prior.
* Ability to read, write and understand English.
* Experienced at least a 25% total weight loss since surgery.
* BMI at least 27 kg/m.
* Weight regain of no more than half of excess body weight. These cases will be referred back to the surgeon.

Exclusion Criteria:

* Taking Weight-suppressing medication (e.g. phentermine, bupropion)
* On medications known to cause weight gain
* Change in smoking status with past three months
* Change in antidepressant or other psychotropic medication or dosage in past six weeks
* Change in psychotherapy status in past six weeks
* Current purging behaviors occurring more than once per week over the past six weeks (vomiting or laxative/diuretic use for the purpose of weight loss
* Current alcohol abuse or dependence or illicit drug use in past three months
* Active bipolar or psychotic spectrum disorder
* Current suicidality or homicidality
* Severe neuropsychological disease (history of seizure, uncontrolled hypertension
* Condition associated with cognitive dysfunction (e.g. Alzheimer's dementia, other neurological conditions)
* Medically unstable condition or one which the investigators feel put the participant at risk in the study
* Functional limitations-not able to walk 2 block without assistance
* Exercise is contra-indicated (e.g., severe cardiovascular disease, uncontrolled hypertension, hematocrit.<30%, chronic kidney disease, severe pulmonary disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-07; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Weight Regain After Bariatric Surgery | 6 months
  The overall goal of the project is to collect pilot data for a RO1 application. The primary outcome will be kg lost and BMI units lost from pre- to post-treatment. The effect size (Mean1 - Mean2 / pooled s.d.) of the intervention will be determined for within subject and between subject differences. It is hypothesized that a moderate effect size (.5) will be demonstrated and that has been selected a priori as the criteria for pursuing a larger-scale randomized clinical trial.

SECONDARY OUTCOMES:
Daily caloric intake | 6 months
  Subjects will keep a food intake diary and bring it to their appointments where calorie intake will be calculated
Daily protein intake | 6 months
  Subjects will keep a food intake diary and bring it to their appointment where daily protein intake will be calculated
Number of minutes of physical activity | 6 months
  Subjects will wear a pedometer to track their daily activity
Presence of disordered eating behaviors | 6 months
  Subjects will complete pre and post treatment questionnaires to assess for disordered eating behaviors

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Heinberg, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States